CLINICAL TRIAL: NCT02987478
Title: Effect of Vitamin D Status on Clinical Pregnancy Rates Following Intra Cytoplasmic Sperm Injection
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ain Shams Maternity Hospital (Other)
Responsible Party: Principal Investigator, Alaa Sayed Abdul-hafeez, Clinical Professor, Ain Shams Maternity Hospital
Other Study IDs: 6789
Record Dates: First submitted 2016-11-29; First posted 2016-12-09 (Estimated); Last update posted 2016-12-09 (Estimated); Status verified 2016-12

CONDITIONS: Infertility
Keywords: Vitamin D following intra cytoplasmic sperm injection
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

SUMMARY:
All patients will undergo in vitro fertilization.

Serum 25 (OH) D samples will be collected within1 week before oocyte retrieval.

Whole blood specimens will be collected in serum separator tubes using acceptable medical techniques to avoid hemolysis.

Ultrasound guided fresh embryo transfer will be performed on day 5 after fertilization.

clinical pregnancy will be confirmed by observation of intrauterine sac visible on ultrasound performed 4-5 weeks after embryo transfer.

DETAILED DESCRIPTION:
PATIENTS AND METHODS

Protocol Outline:

The Study:

Study site:

Ain Shams University Maternity Hospital.

Study Design:

A prospective Cohort study.

Study setting:

The study will be conducted at Ain Shams University Maternity Hospital.

Study population:

The study will include all women planned to undergo IVF due to unexplained infertility.

Methodology:

The study will be approved by the hospital ethics committee.

All included women will undergo the following:

* History taking.
* General and abdominal examination.
* Vaginal examination and assessment
* Pelvic ultrasound.
* Routine laboratory investigations including complete blood picture, hematocrit, liver and kidney function tests and coagulation profile.
* Preoperative senior anesthetist assessment.
* Hysteroscopy.

All patients will undergo IVF.

Serum 25(OH)D samples will be collected within1 week before oocyte retrieval.

Whole blood specimens will be collected in serum separator tubes using acceptable medical techniques to avoid hemolysis.

Ultrasound-guided fresh embryo transfer will be performed on day 5 after fertilization.

clinical pregnancy will be confirmed by observation of intrauterine sac visible on ultrasound performed 4-5 weeks after embryo transfer.

Measurement of Outcomes

1. serum 25 (OH) D levels.
2. Number of oocyte.

   Most studies put the optimal number of retrieved oocytes between 10 and 15.
3. The implantation rate:

   Calculated as the number of gestational sacs observed by ultrasound divided by the number of embryos transferred, multiplied by 100.
4. Number of gestational sac.

ELIGIBILITY:
Inclusion Criteria:

* Age between 20 and 35 years old.
* Body mass index between 20 - 30.
* Unexplained infertility .
* Follicle-stimulating hormone level 12 IU/L or lower (baseline level, cycle day 3).
* Normal hysteroscopy ( healthy uterus with no fibroids or other growths)
* Fresh embryo transfer of 2 or more blastocysts stage.
* Embryo transfer on day 5 after fertilization

Exclusion Criteria:

* Women younger than 20 years old or older than 35 years old.
* Previous one or more failed IVF.
* Uncorrected congenital or acquired uterine anomalies.
* Other causes of infertility rather than unexplained infertility.
* Less than 2 embryo transfer, cleavage stager frozen embryo transfer.

Ages: 20 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Age between 20 and 35 years old.
  * Body mass index between 20 - 30.
  * Unexplained infertility .
  * Follicle-stimulating hormone level 12 IU/L or lower (baseline level, cycle day 3).
  * Normal hysteroscopy .
  * Fresh embryo transfer of 2 or more blastocysts stage.
  * Embryo transfer on day 5 after fertilization
Sampling Method: Probability Sample
Enrollment: 240 (Estimated)
Dates: Start 2016-03; Primary Completion 2017-03 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
pregnancy | 4-5 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University Maternity Hospital, Cairo, Abbassia, Egypt